CLINICAL TRIAL: NCT02530333
Title: Differential Biomechanical Effects of an ACL Injury Prevention Program in Women's Basketball and Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: High Point University (Other)
Collaborators: University of North Carolina, Greensboro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201404-370
Record Dates: First submitted 2015-05-21; First posted 2015-08-21 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Basketball Control (No Intervention): Control group of basketball players
- Basketball intervention (Experimental): Intervention group of basketball players
  Interventions: Other: Neuromuscular Prevention Program
- Soccer Control (No Intervention): Control group of soccer players
- Soccer Intervention (Experimental): intervention group of soccer players
  Interventions: Other: Neuromuscular Prevention Program

INTERVENTIONS:
Other: Neuromuscular Prevention Program — Participants in the intervention group will complete at 6 week ACL injury prevention program previously described in the literature as being effective at reducing ACL injury risk. The prevention program lasts 20-25 minutes in duration and will take place as a warm-up prior to any practice. The frequency will depend solely on the number of practices each team holds throughout the given 6-week time period.
  Arms: Basketball intervention; Soccer Intervention

SUMMARY:
Anterior cruciate ligament injury programs are less successful in women's basketball than soccer players, yet the reason for this discrepancy is unknown. Thus, this study will recruit high school aged girl's basketball and soccer players, randomized teams into control and experimental groups, administer an ACL injury prevention program in the experimental group and compare the two groups on their lower extremity biomechanics before and after completion of the program. Biomechanical analyses will help determine the extent to which women's basketball and soccer players respond differently to a uniform injury prevention program, and whether this prevention program provides an adequate stimulus to improve lower extremity biomechanics during basketball-specific tasks.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injury prevention programs are considerably less successful in women's basketball than women's soccer. Women's basketball and soccer are each characterized by distinct sport-specific demands, where women's basketball players perform significantly more frequent jumping (2- and 1-legged landings) and frontal plane movements than women's soccer players. Despite varying sport-specific demands, ACL injury prevention programs have been uniformly administered in both sports, and emphasize improving high-risk biomechanics during 2-legged sagittal plane tasks. As such, they may not provide the appropriate stimulus to reduce ACL injury risk during the high-risk demands associated with women's basketball. To date, the differential biomechanical adaptations that result from ACL injury prevention programs in women's basketball and soccer have never been investigated.

This study will use a cluster randomized controlled trial using a repeated measures design. Participants will be randomized (by team) in to control and intervention groups. Participants in the control group will be asked to continue their normal daily and athletic activities (practices, games) without participating any distinct injury prevention training. Participants in the intervention group will complete at 6 week ACL injury prevention program previously described in the literature as being effective at reducing ACL injury risk. The prevention program lasts 20-25 minutes in duration and will take place as a warm-up prior to any practice. The frequency will depend solely on the number of practices each team holds throughout the given 6-week time period. A member of the research team plans to be at each intervention session. All participants will complete pre- and post-testing approximately 1 week before the onset and after the completion of the prevention program, respectively. As stated previously, all pre- and post-testing will be performed at the High Point University Human Biomechanics and Physiology Laboratory.

The following are Specific Aims and Hypotheses. Specific Aim 1. To determine the extent to which women's basketball and soccer players employ distinct lower extremity movement strategies during sagittal and frontal plane jump landing tasks.

Hypothesis 1. Prior to training, women's basketball athletes will exhibit no significant differences in high-risk hip and knee kinematics, but will generate higher hip and knee joint moments during jump landing activities than women's soccer players.

Specific Aim 2. To determine the response of women's basketball and soccer athletes to a 6-week ACL injury prevention program, as measured by changes in multi-planar hip and knee biomechanics of jump landings during sagittal and frontal plane jump landing tasks.

Hypothesis 1. After 6 weeks of training, high-risk biomechanics will improve to a larger extent during sagittal plane than frontal plane jump landing tasks.

Hypothesis 2. After 6 weeks of training, there will be no significant differences in biomechanical changes in women's basketball compared to women's soccer players.

ELIGIBILITY:
Inclusion Criteria:

* Participants will need to be participating in high school aged, competitive-level basketball and/or soccer and are medically cleared to participate in sports.

Exclusion Criteria:

* Participants will be excluded if they have a history of lower extremity surgery in the past 6 months, or have been diagnosed with a vestibular, balance, or cardiovascular disorders that may preclude safe participation during landing and jumping activities.

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Angular Kinematics (hip flexion, hip adduction, hip internal rotation, knee flexion, abduction, knee internal rotation, knee external rotation) | 6-8 weeks
Lower Extremity Kinetics (hip flexion, hip adduction, hip internal rotation, knee flexion, abduction, knee internal rotation, knee external rotation external moments) | 6-8 weeks

SECONDARY OUTCOMES:
Triple Jump Distance | 6-8 weeks
Maximal Vertical Jump Height | 6-8 weeks
  Countermovement jump
Agility | 6-8 weeks
  T-test

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Taylor, DPT, Principal Investigator — High Point University
Locations (1):
- High Point University, High Point, North Carolina, United States

REFERENCES:
- [Derived] Taylor JB, Nguyen AD, Shultz SJ, Ford KR. Hip biomechanics differ in responders and non-responders to an ACL injury prevention program. Knee Surg Sports Traumatol Arthrosc. 2020 Apr;28(4):1236-1245. doi: 10.1007/s00167-018-5158-1. Epub 2018 Sep 27. PMID 30259145
- [Derived] Taylor JB, Ford KR, Schmitz RJ, Ross SE, Ackerman TA, Shultz SJ. Sport-specific biomechanical responses to an ACL injury prevention programme: A randomised controlled trial. J Sports Sci. 2018 Nov;36(21):2492-2501. doi: 10.1080/02640414.2018.1465723. Epub 2018 Apr 19. PMID 29671383